CLINICAL TRIAL: NCT00919282
Title: A Multi Center Phase II Study of 5-Fluorouracil/ Folinic Acid Plus Gemcitabine in Patients With Advanced Pancreatic Cancer.
Brief Title: Gemcitabine (GFF) in Patients With Pancreatic Cancer
Acronym: GFF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CONKO-Studiengruppe (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: CONKO-Studiengruppe, Universitätsmedizin Berlin
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONKO 002 pilot
Record Dates: First submitted 2009-06-09; First posted 2009-06-12 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; gemcitabine; combination
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine/folinic acid/5-FU (Experimental): Gemcitabine 1g/m² 5-FU 750mg/m² FS 500 mg/m²
  Interventions: Drug: gemcitabine, folinic acid, 5-FU

INTERVENTIONS:
Drug: gemcitabine, folinic acid, 5-FU — gemcitabine 1g/m² - 30 minutes folinic acid 500mg/m² - 2 hours 5-FU 750mg/m² - over 24hours
  Other Names: gemzar; oncofolic; 5-fu

SUMMARY:
The purpose of this study is to examine the efficacy and safety of the drug combination GFF in patients with advanced pancreatic cancer (APC).

DETAILED DESCRIPTION:
This open-label, multi center phase II study was conducted to investigate the efficacy and safety of the combination of 5-Fluorouracil (5-FU)/folinic acid (FA) plus gemcitabine (GFF) in patients (pts) with advanced pancreatic cancer (APC). We consequently started this study after completing the phase I trial accomplished by our CONKO- study group.

ELIGIBILITY:
Inclusion Criteria:

* histological proved pancreatic cancer
* inoperable disease
* informed consent
* adequate bone marrow reserve

Exclusion Criteria:

* under 18 years
* brain metastasis
* lactating woman
* life expectancy under 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 1997-09; Primary Completion 2000-07 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 1 year

SECONDARY OUTCOMES:
safety of treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: helmut oettle, MD, Principal Investigator — CONKO-Studiengruppe
Locations (1):
- Universitätsmedizin Berlin, Berlin, State of Berlin, Germany